CLINICAL TRIAL: NCT00660101
Title: OVax®: A Feasibility Study Using a DNP-Modified Autologous Ovarian Tumor Cell Vaccine as Therapy in Ovarian Cancer Patients After Relapse:
Brief Title: Trial of Autologous, Hapten-Modified Vaccine, OVAX, in Patients With Relapsed Stage III or IV Ovarian Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AVAX Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A/100/0501
Record Dates: First submitted 2008-04-16; First posted 2008-04-17 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Adenocarcinoma of the Ovary
Keywords: ovarian cancer; vaccine; immunotherapy; autologous
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 5 million OVax: Autologous, DNP-Modified Ovarian Cancer Vaccine cells
  Interventions: Biological: OVax: Autologous, DNP-Modified Ovarian Cancer Vaccine
- 2 (Experimental): 2.5 million OVax: Autologous, DNP-Modified Ovarian Cancer Vaccine cells
  Interventions: Biological: OVax: Autologous, DNP-Modified Ovarian Cancer Vaccine
- 3 (Experimental): 0.5 million OVax: Autologous, DNP-Modified Ovarian Cancer Vaccine cells
  Interventions: Biological: OVax: Autologous, DNP-Modified Ovarian Cancer Vaccine

INTERVENTIONS:
Biological: OVax: Autologous, DNP-Modified Ovarian Cancer Vaccine — OVax: Autologous, DNP-Modified Ovarian Cancer Vaccine cells in suspension dosage - depends on arm route - intradermal frequency - weekly x7, booster at 6 months
  Other Names: OVax; O-Vax

SUMMARY:
To determine if a vaccine made from the patient's own tumor tissue can stimulate an immune response against the patient's tumor cells. To determine the safety of the vaccine.

DETAILED DESCRIPTION:
To study the toxicity, safety and DTH response of DNP-modified autologous ovarian tumor cell vaccine and the DTH response to unmodified ovarian tumor cells in patients with relapsed ovarian cancer:

* To determine the tolerability and toxicity of the treatment regimen
* To determine whether O-Vax induces a DTH response to autologous, DNP-modified ovarian cancer cells
* To determine whether O-Vax induces a DTH response to autologous, unmodified ovarian cancer cells

Study Population: Patients with recurrent epithelial ovarian cancer whose therapeutic tumor surgery provides a mass which yields adequate tumor cells for vaccine preparation and delayed-type hypersensitivity (DTH) testing

Study Design: A Phase I/IIa double-blind, three-dose, multi-center study

Investigational Product: O-Vax: DNP-modified autologous ovarian tumor cell vaccine

Dosage Form: Cell suspension

Route of Administration: Intradermal

Dosage and Treatment Schedule: Prior to enrollment in the study, one dose of 5 x 106 modified and one dose of 5 x 106 unmodified autologous ovarian cancer cells will be administered, to establish a negative DTH response at baseline. Three dosing regimens will be used: 5 x 105, 2.5 x 106, or 5 x 106 DNP-modified autologous ovarian tumor cells. An initial dose of DNP-modified autologous ovarian tumor cells* followed by cyclophosphamide then weekly doses of DNP-modified autologous ovarian tumor cells mixed with Bacillus of Calmette and Guérin (BCG) for 6 weeks, and completed with one dose of DNP-modified autologous ovarian tumor cells mixed with BCG as a 6 month booster if adequate cells

* count determined prior to aliquoting for cryopreservation

Endpoints: Treatment-emergent and related adverse events, serious adverse events, and Grade 3 and 4 laboratory abnormalities

Other Parameters:

* Delayed-type hypersensitivity skin reactions for assessing the induction of immune responses to DNP-modified and unmodified autologous ovarian tumor cells
* CA-125 levels
* Survival
* Exploratory analysis incorporating in vitro analysis of lymphocytes separated from patient blood samples

Duration of Treatment: Up to 6 months

Duration of Subject Participation in Study: Three months from the patient's last vaccine

Duration of Follow-up: Survival information will be collected via phone or visit on a quarterly basis for each patient beginning 30 days after the last scheduled visit

Number of Subjects Required to Meet Protocol Objectives: 42 evaluable subjects

Number of Study Centers: 4-5

Number of Individual Blood Draws: 13 draws over nine months

Volume of Blood Drawn: 11 Draws of 30 mL/draw (total 360 mL) and two draws of 50mL in heparinized tubes

ELIGIBILITY:
Inclusion Criteria:

Screening Phase

* Stage III or IV adenocarcinoma of ovary
* Candidate for surgery to excise the tumor
* Signed informed consent for tumor acquisition

Treatment Phase

* At least 18 years of age
* Standard surgical debulking to maximum extent possible
* Adequate amount of tumor tissue obtained from surgical debulking to prepare a series of vaccines and skin test materials.
* Administration of intraperitoneal chemotherapy following surgical debulking Intraperitoneal drug to consist of a taxane (paclitaxel or docetaxel) Dose of taxane: paclitaxel=60-75 mg/m2 / weekly x 4 or docetaxel = 25 mg/m2 - weekly x 4
* Vaccines and DTH materials pass lot release
* Minimum of 2 weeks and maximum of 6 weeks following last dose of intraperitoneal chemotherapy
* Immunocompetent, as determined by anergy panel performed 1 week after last dose of intraperitoneal chemotherapy (baseline PPD+ patients allowed)
* Expected survival of at least 6 months
* Karnofsky performance status ³ 80
* Signed informed consent for protocol participation

Exclusion Criteria:

* Alkaline phosphatase > 2.5 x ULN
* Total bilirubin > 2.0 mg/dL
* Creatinine > 2.0 mg/dL
* Hemoglobin < 10.0 g/dL
* WBC < 3,000 /mm3
* Platelet count < 100,000/mm3
* Major field radiotherapy within 6 months prior to participation in the study
* Brain metastases, unless successfully treated at least 6 months prior to entry
* Prior immunotherapy (interferons, tumor necrosis factor, other cytokines [e.g., interleukins], biological response modifiers, or monoclonal antibodies) within 4 weeks prior to participation in the study
* Prior splenectomy
* Concurrent use of systemic steroids (Note: Topical steroid therapies [applied to the skin] are not contraindicated for participation in the study, provided these are not applied to either arm. Inhaled aerosol steroids are not contraindicated for participation in the study.)
* Concurrent use of immunosuppressive drugs
* Concurrent use of antitubercular drugs (isoniazid, rifampin, streptomycin)
* Other malignancy within 5 years except curatively treated non-melanomatous skin cancer and curatively treated carcinoma in situ of the uterine cervix
* Concurrent autoimmune diseases, e.g., systemic lupus erythematosus, multiple sclerosis or ankylosing spondylitis
* Concurrent medical condition that would preclude compliance or immunologic response to study treatment
* Concurrent serious infection or other serious medical condition
* Receipt of any investigational medication within 4 weeks prior to participation in the study
* Known gentamicin sensitivity
* Anergic, defined by the inability to make a DTH to at least one of the following: candida, mumps, tetanus, trichophyton (based upon availability), or PPD
* Vaccine lot release failure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Cell-mediated immunity to autologous tumor cells | 3 months

SECONDARY OUTCOMES:
Safety | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Henry E Schea, Study Director — AVAX Technologies
Locations (3):
- United States (3):
  - Cancer Treatment Centers of America (CTCA-Midwestern), Zion, Illinois
  - Cancer Treatment Centers of America (CTCA-Southwestern), Tulsa, Oklahoma
  - Cancer Treatment Centers of America (ERMC), Philadelphia, Pennsylvania

REFERENCES:
- [Background] Dunton CJ, Carlson JA, King SA, Bloome E, Neufeld J, Berd D. Immunological and clinical effects of autologous hapten-modified vaccine in patients with advanced ovarian carcinoma., 19: Abstract 1828 ed 2000. p. 466a.
- [Background] Berd D, Sato T, Maguire HC Jr, Kairys J, Mastrangelo MJ. Immunopharmacologic analysis of an autologous, hapten-modified human melanoma vaccine. J Clin Oncol. 2004 Feb 1;22(3):403-15. doi: 10.1200/JCO.2004.06.043. Epub 2003 Dec 22. PMID 14691123
- See also: AVAX Technologies — http://www.avax-tech.com
- See also: Cancer Treatment Centers of America — http://www.cancercenter.com